CLINICAL TRIAL: NCT01386268
Title: KOGENATE® FS , Local Post Authorization Safety Study
Brief Title: Kogenate FS Regulatory Post-Marketing Surveillance
Acronym: KG0910KR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14927; KG0910KR (Other: Company Internal)
Record Dates: First submitted 2011-06-14; First posted 2011-07-01 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Hemophilia A
Keywords: Kogenate FS; Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Patients with diagnosis of hemophilia A, treated with KOGENATE FS as their only source of FVIII, decision taken by the investigator to administer KOGENATE FS

SUMMARY:
To obtain data on safety, efficacy, and tolerability of KOGENATE FS under real-life conditions in its registered indications.

The observation period for each patient is up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of hemophilia A
* Treated with KOGENATE FS as their only source of FVIII, decision taken by the investigator to administer KOGENATE FS
* Signed the informed consent form to participate in this study.
* For pretreated patients with more than 100 exposure days an inhibitor assessment within three months prior to enrollment should be available
* For pretreated patients with less than 100 exposure days an inhibitor assessment at baseline should be available
* For patients with no available inhibitor status, it should be checked as per the recommendation of KFDA
* Patients are defined as included in the study if there is a documented prescription of KOGENATE FS by the physician.

Exclusion Criteria:

* Patients with hypersensitivity to any ingredient of KOGENATE FS or to the protein of mouse or hamster will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia A in Korea
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | Up to 6 months

SECONDARY OUTCOMES:
Type of the treatment (prophylaxis, on demand, surgery) | Initial visit and 6 month f/u or at the end of the observation visit
Total consumption of FVIII | Initial visit and 6 month f/u or at the end of the observation visit
Daily dosage/frequency of FVIII (if used for prophylaxis, on demand, surgery/peri-operatively) | Initial visit, 6 month follow-up visit and 12 month follow-up visit
General assessment of therapy by physician by grading from 1 to 4: 1) excellent; 2) good; 3) sufficient; 4) insufficient | 6 month f/u or at the end of observation visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea